CLINICAL TRIAL: NCT06712095
Title: Video Capsule Examination in Patients With Lynch and Other Cancer-predisposition Syndromes - a Proof-of-concept Study for Obtaining Data to Support the Development of Machine Learning Algorithms to Detect Early Cancers
Brief Title: Video Capsule Examination in Patients With Lynch Syndrome
Acronym: PILLCAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CCR5717
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Lynch Syndrome; Li Fraumeni Syndrome; PTEN Hamartoma Syndrome; FAP; MUTYH Biallelic Mutation; STK11 Mutation; CDH1 Gene Mutation; CHEK2 Gene Mutation; BMPR1A Gene Mutation; SMAD4 Gene Mutation
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis; Li-Fraumeni Syndrome; Hamartoma Syndrome, Multiple | interventions — Physical Examination; Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Videocapsule investigation (Experimental)
  Interventions: Device: Video capsule investigation

INTERVENTIONS:
Device: Video capsule investigation — Participants will undergo both a video capsule examination and a colonoscopy on the same day.
  Other Names: Colonoscopy

SUMMARY:
Surveillance for colorectal cancer (CRC) in patients predisposed to develop CRC during their lifetime has been impacted by access to colonoscopy suites and endoscopy specialists in the past couple of years. An alternative method, namely the colon capsule, has been proposed, however this investigation is time consuming for the clinician and the images require up to one hour (30-60 minutes) reading to issue a result. The investigators propose to obtain images from paired colonoscopies and colon capsules with the purpose of developing an AI algorithm which could aid the clinicians in reading the colon and expand access to this investigation.

The main aim of the study is to determine whether it is possible to obtain usable paired images from patients with Lynch and other cancer predisposition syndromes. This will depend on the willingness of the patients to take part in the study and the technical ability of obtaining data from paired images of colonoscopies and colon capsule.

At recruitment, participants will undergo a colon capsule investigation, followed by a routine colonoscopy as per their normal standard of care. Paired endoscopic images from colonoscopies and colon capsules will be collected and anonymised data will be accessed by the bioinformatician for analysis.

If the study will be successful in reaching the primary endpoint, further trials will be opened, allowing for a larger population to be included and to obtain more robust data, which eventually can lead to validated AI algorithms and application of computer-aided video-capsules examination as a screening tool in at-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 years old with no active cancer
* No previous resection of the colon and/or rectum
* Carriers of a pathogenic/likely pathogenic variant in any of the following cancer-predisposition genes: Lynch syndrome (MLH1, MSH2, MSH6, PMS2), APC (FAP syndrome); biallelic MUTYH; STK11 (Peutz-Jeghers syndrome); PTEN, CDH1, CHEK2, TP53, BMPR1A and SMAD4 (Juvenile polyposis syndrome)
* Able to consent to the study and undergo colonoscopy.

Exclusion Criteria:

* Extensive surgery which poses a high risk of video-capsule blockage or narrowing of the bowel due to extensive tumour. Extensive surgery implies any removal of large portions of the small or large bowel that might cause a narrowing (stricture) in the digestive tract.
* Previous irradiation to abdomen or pelvis (risk for small bowel obstruction)
* Carriers of a variant associated with reduced penetrance (in the view of a geneticist) or a variant of uncertain significance.
* Patients with a PS of 3 or 4 and/or mobility issues
* Pregnancy
* Pacemaker or internal electro-medical device (artificial heart valve, cochlear implant or an internal electromedical device).
* Insulin-dependent diabetes
* Patients who require deep sedation for colonoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of paired images the bioinformatician assesses as useful for the development of algorithm | 18 months

SECONDARY OUTCOMES:
The proportion of patients at high-risk as defined by inclusion criteria who agree to undergo video capsule examination. | 18 months
The proportion of patients who undergo both video capsule examination and colonoscopy, from whom it is possible to obtain paired images | 18 months
The description of any adverse events collected for the Pillcam procedure. | 18 months
  All adverse events will be collected using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lee, PhD, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- The Royal Marsden NHS Foundation Trust, London, (Select), United Kingdom